CLINICAL TRIAL: NCT07171554
Title: Clinical Performance Study of a New Diagnostic Test for Drug Sensitivity Evaluation in Metastatic Colorectal Cancer
Brief Title: Evaluation of a Diagnostic Test to Identify the Best Drugs for Treatment of Metastatic Colorectal Cancer
Acronym: DSEE-CRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncosyne AS (Industry)
Collaborators: University Hospital, Akershus (Other); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DSEE-CRC; 2024-519600-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-20; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: patient-derived tumoroids; in vitro diagnostics; drug screening; clinical performance study; randomized; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- µCAN guided therapy (Experimental): The treating physician may use the µCAN diagnostic drug screen report to guide therapy
  Interventions: Diagnostic Test: µCAN drug screen test
- Standard-of-Care (Other): The patient will be given the Standard-of-Care in the 3rd line setting, trifluridine/tipiracil/bevacizumab
  Interventions: Other: Standard-of-Care Therapy

INTERVENTIONS:
Diagnostic Test: µCAN drug screen test — µCAN guided therapy is based on drug screening of patient-derived tumoroids. The patient might be treated with clinically relevant on-label or off-label drugs
  Arms: µCAN guided therapy
Other: Standard-of-Care Therapy — trifluridine/tipiracil/bevacizumab combination, 28 day cycles
  Arms: Standard-of-Care

SUMMARY:
DSEE-CRC is a top-tier Norwegian and Swedish public-private partnership for the development of µCAN, a unique patient-centric, therapy-guiding in vitro diagnostic test to improve cancer treatment outcomes for metastatic colorectal cancer patients. µCAN takes a cancer biopsy sample as input and combines proprietary patient-derived tumoroid culturing conditions with state of-the-art machine learning, and computer-vision guided fluorescence high- content drug screening and analysis, to identify the best therapeutical approach for clinical practice. DSEE-CRC will have a positive societal and financial impact and directly contributes to the Good Health and Well-being Sustainable Development Goals by delivering patient-tailored treatments, concurrently increasing cancer survivability rates, improving patients' quality of care, and reducing cancer treatment costs for healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent (for each part of the study) for participation in the clinical performance study.
* Male or female patients, ≥18 years of age, with Eastern Cooperative Oncology Group (ECOG) performance status 0-1, who have metastatic lesions in the liver or peritoneum (or lymph nodes) that are radiologically assessable and can be biopsied, and who have recently failed 1st line systemic therapy (2nd line for patients with three standard therapy lines) for unresectable metastatic disease and will shortly commence a new line of standard therapy.
* Patient is eligible for another line of tumour directed therapy on failure of the SoC.
* Patient has the following laboratory values, as measured in serum/plasma within 14 days prior to signing of informed consent for participation in Part A and B, respectively, indicative of adequate organ function:

  * Haemoglobin at least 10.0 g/dL.
  * Neutrophils at least 1.5 x109/L (without current use of colony-stimulating factors).
  * Platelets at least 100 x109/L.
  * AST/ALT no higher than 2xULN when patient does not have metastatic disease in the liver, or no higher than 5xULN when patient has metastatic disease in the liver.
  * Bilirubin no higher than 1.5xULN when patient does not have metastatic disease in the liver, or no higher than 2xULN when patient has metastatic disease in the liver.
  * Albumin no lower than 30 g/L.
  * INR within normal level.
  * Creatinine no higher than 1.5xULN.
* For Part A: the treating physician should follow contraceptive requirements described in the SmPC of respective treatment.
* For Part B: women of childbearing potential (WOCBP) must practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the patient) or must agree to use a highly effective method of contraception with a failure rate of <1 % to prevent pregnancy from at least 2 weeks prior to the screening visit of Part B to 4 weeks after the last administration of IMP in Part B. In addition, any male partner of a female participant must, unless he has undergone vasectomy, agree to use a condom from the screening visit of Part B until 4 weeks after the last administration of IMP in Part B.

The following are considered highly effective methods of contraception:

* combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
* progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable),
* intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) WOCBP must refrain from donating eggs from the first IMP administration until 3 months after the last IMP administration. WOCBP with an exclusive male partner who has undergone vasectomy may chose not to use contraceptives.

Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] >25 IU/L is confirmatory). Male participants must be willing to use condom or be vasectomised or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the first administration of IMP until 4 weeks after the last administration of IMP. Any female partner of a non-vasectomised male participant who is of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to the first administration of IMP to 4 weeks after the last administration of IMP.

Exclusion Criteria:

* Life expectancy < 3 months.
* Planned treatment or treatment with another investigational drug or investigational device within 3 months prior to the day of the tumour sampling procedure.
* Patients who are pregnant, or currently breastfeeding.
* Investigator considers the patient unlikely to comply with clinical performance study procedures, restrictions and requirements.
* Part B only: no µCAN report was generated from Part A.
* Part B only: Patient is not eligible for trifluridine/tipiracil/bevacizumab combination therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a successful biopsy yielding a µCAN report. | Through completion of study Part A, an average of 6 months
  To evaluate the performance of µCAN to generate high-quality, accurate, robust and reliable data intended as guidance in the physician's choice for 3rd line therapy for patients with mCRC (Part A)

SECONDARY OUTCOMES:
Proportion of patients with a successful biopsy yielding a µCAN report within 56 days (8 weeks). | Through completion of study Part A, an average of 6 months
  To evaluate the performance of µCAN to generate high-quality, accurate, robust and reliable data intended as guidance in the physician's choice for 3rd line therapy for patients with mCRC (Part A)
Proportion of patients with a successful biopsy yielding a µCAN report with at least one drug therapy nomination. | Through completion of study Part A, an average of 6 months
  To evaluate the performance of µCAN to generate high-quality, accurate, robust and reliable data intended as guidance in the physician's choice for 3rd line therapy for patients with mCRC (Part A).
Frequency, intensity and seriousness of adverse events (AEs) related to device or study procedures. | Through completion of study Part A, an average of 6 months
  To demonstrate compliance with the general safety and performance requirements for µCAN (Part A).
Frequency and nature of device deficiencies (DD). | Through completion of study Part A, an average of 6 months
  To demonstrate compliance with the general safety and performance requirements for µCAN (Part A).

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Ree, MD, Professor of Oncology, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No